CLINICAL TRIAL: NCT06155708
Title: Exogenous Ketone Supplementation to Improve Cardiovascular Disease Risk Factors in Females with Polycystic Ovary Syndrome
Brief Title: Exogenous Ketone Supplementation in Females with Polycystic Ovary Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Charlotte Usselman, Primary Investigator, McGill University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-9710
Record Dates: First submitted 2023-10-18; First posted 2023-12-04 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: PCOS
Keywords: Polycystic ovary syndrome; Ketone monoester ingestion; Insulin resistance; Endothelial function; Blood pressure; Oral glucose tolerance test; Flow mediated dilation; Handgrip exercise; Neurovascular transduction; Cold pressor test
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Ketones; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone (Experimental): - Ketone monoester supplement in the form of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.45ml/kg body weight) ingested with water and vanilla-flavored stevia in a total volume of 100 ml.
  Interventions: Dietary Supplement: Ketone
- Placebo (Placebo Comparator): 100 ml water combined with 10ml bitter flavor and vanilla-flavored stevia
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Ketone — - Ketone monoester supplement in the form of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.45ml/kg body weight) ingested with water and vanilla-flavored stevia in a total volume of 100 ml.
  Arms: Ketone
Dietary Supplement: Water — 100 ml water combined with 10ml bitter flavor and vanilla-flavored stevia
  Arms: Placebo

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 1 in 5 females of reproductive age. Commonly characterized as a disorder of infertility, PCOS is often accompanied by 3 potent cardiovascular disease (CVD) risk factors: insulin resistance, endothelial dysfunction, and elevated blood pressure. Accordingly, PCOS is associated with the development of CVD, the second leading cause of death in females in Canada. However, effective treatments to improve cardiovascular health in PCOS are lacking.

Exogenous ketone monoester (KME) ingestion has been shown to improves outcomes associated with insulin resistance, endothelial function, and blood pressure regulation in healthy individuals and individuals predisposed to CVD. Therefore, oral ketone supplements offer a practical and effective strategy for improving cardiovascular health; however, this treatment has yet to be evaluated in PCOS.

Therefore, the overall goal of this project is to employ KME ingestion to improve markers of cardiovascular health in females with PCOS.

On two different days, participants will consume either a beverage containing a ketone supplement or a beverage containing a placebo supplement. The objectives are to compare responses between KME and placebo ingestion, and examine all outcomes related to cardiovascular health in females with PCOS in comparison with female controls of similar age and body mass index. The effects of KME ingestion will be quantified on: 1) glycemic control during an oral glucose tolerance test; 2) endothelial function using the flow-mediated dilation test; 3) blood pressure and acute blood pressure regulation; and 4) hemodynamic responses to acute exercise.

ELIGIBILITY:
Inclusion Criteria:

* All female participants will report female sex assigned at birth
* All participants will be aged 18 to 40
* PCOS diagnosis

Exclusion Criteria:

* Current smokers or a prolonged history of smoking
* Presence or history of overt cardiometabolic disease (e.g., stage 2 hypertension, diabetes, heart disease), neurologic disease, or endocrinopathy (with the exception of PCOS)
* Current pregnancy or currently breastfeeding
* Current use of medications which may affect our outcomes of interest (e.g., anti-hypertensives, anti-androgens, metformin)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic responses to a 2-hr oral glucose tolerance test | 0-2.5 hours in the post-prandial period
  - Glucose is calculated by the area under the curve using the trapezoid method.
Flow mediated dilation (FMD) | 30 minutes
  - Endothelial function is assessed using the standard FMD; quantified as the percent increase in diameter from rest to peak diameter observed during reactive hyperemia (%FMD). The % change in diameter reflects the ability of the vessel to dilate in response to sheer stress induced by the flow following the release of occlusion. This reflects the function of the endothelium, or release of nitric oxide.
Systolic Blood Pressure (SBP) | 2 hours
  - SBP, measured in mmHg
Diastolic Blood Pressure (DBP) | 2 hours
  - DBP, measured in mmHg

SECONDARY OUTCOMES:
Insulin area under the curve | 0-2.5 hours in the post-prandial period
  - Insulin area under the curve during oral glucose tolerance test
C-peptide | 0-2.5 hours in the post-prandial period
  - C-peptide area under the curve during oral glucose tolerance test
Glucagon-like peptide-1 (GLP-1) | 0-2.5 hours in the post-prandial period
  - GLP-1 area under the curve during oral glucose tolerance test.
Glucose-dependent insulinotropic polypeptide (GIP) | 0-2.5 hours in the post-prandial period
  - GIP area under the curve during oral glucose tolerance test.
Triglycerides | 0-2.5 hours in the post-prandial period
  - Triglycerides area under the curve during oral glucose tolerance test
Insulinogenic index | 0-2.5 hours in the post-prandial period
  - (Insulin at 30 min - fasting insulin)/ (plasma glucose at 30 min- fasting plasma glucose).
Arterial artery blood flow | 0-2.5 hours in the post-prandial period
  - Calculated as the product of mean blood flow velocity (cm/sec) and cross-sectional area (2Πr2) x 60 sec/min.
Shear rate and low-flow mediated vasoconstriction to the FMD | 30 minutes
  - Shear rate calculated as area under the curve from cuff deflation to the time of peak dilation using the trapezoidal rule, as well as low flow-mediated vasoconstriction during forearm occlusion, which provides an index of the endothelial contribution to resting vascular tone and which predicts cardiovascular disease risk.
Muscle sympathetic nerve activity (MSNA) | 2 hours
  - Measured using microneurography, and expressed in burst/min or bursts/100 heart beats
Neurovascular transduction | 2 hours
  - Assessed by the MSNA signal (recorded in both raw and filtered/rectified/integrated formats for subsequent analyses) and arterial blood flow extracted on a beat-by-beat basis and processed using custom transduction software.
Vascular resistance | 2 hours
  - Calculated as mean arterial pressure divided by Finometer-derived cardiac output
Capillary blood Beta-OHB concentrations | 0-2.5 hours in the post-prandial period
  - Measures in mmol/L
Serum testosterone | 5 minutes
  - Measured in pg/ml.
Serum sex hormone binding globulin | 5 minutes
  - Measured in pg/ml.
Serum estradiol | 5 minutes
  - Measured in pg/ml.
Serum Progesterone | 5 minutes
  - Measured in pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Usselman, Ph.D, Principal Investigator — McGill University
Locations (1):
- Cardiovascular Health and Autonomic Research Laboratory, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No